CLINICAL TRIAL: NCT05756400
Title: Polypharmacy and Associated Risk Factors and Clinical Outcomes for Internal Medicine Patients Discharged From Hospital
Brief Title: Polypharmacy Among Internal Medicine Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Iceland (Other)
Responsible Party: Sponsor
Other Study IDs: UI-2022-Polypharmacy-medicine
Record Dates: First submitted 2023-01-26; First posted 2023-03-06 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-01

CONDITIONS: Internal Medicine
Keywords: Polypharmacy; Potentially Inappropriate Medication List; Risk Factors; Cinical Outcomes; Predication on Medication Related Harm; Discharge; Inappropriate Prescribing; Drug-related side effects and adverse reaction,; Readmisson; Patient discharge; Prediction tool; Start and stop; Beers
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The World Health Organisation Patient Safety Challenge: Medication Without Harm has brought our attention to the importance of medication-related harm as a global public health issue. One of the major contributing factors is polypharmacy, the usage of multiple medicines at the same time. People are getting older and living longer with chronic diseases; they need more medications, which frequently leads to polypharmacy. Subsequently, they are at more risk of medication-related harm. The planned project is an epidemiological study on polypharmacy, medication appropriateness, risk factors, and clinical outcomes post-discharge from a hospital for internal medicine patients.

The study group hypothesise that pre- and post-admission polypharmacy and potentially inappropriate prescribing is common, especially among older patients, patients with a high comorbidity and frailty burden. Our hypothesis is additionally that preadmission polypharmacy and potentially inappropriate prescribing is associated with higher short- and long-term mortality, a longer primary hospitalization length of stay, and a higher risk of readmission.

DETAILED DESCRIPTION:
This is an observational, retrospective, single-centered study using clinical data from the patient's medical record from the hospital, the national prescription database of the Directorate of Health, and the ICD-10 codes from primary care records. For this analysis, medicines will be classified into drug classes based on the first five characters of their WHO Anatomical Therapeutic Chemical (ATC) code. The prevalence (pre) and incidence (post) of polypharmacy (≥5 or more regular medicines) and hyper-polypharmacy (≥10 regular medicines) will be calculated. Potentially inappropriate prescribing will be assessed in individuals ≥65 years, applying Beers 2019, Start and Stopp 2014, explicit prescribing criteria. The analysis will be restricted to older individuals, as Beers criteria have not been validated in younger age groups. The anticholinergic burden will be assessed for all individuals ≥18 years will be assessed by applying the anticholinergic burden scale, and the PRIME tool will be applied to predict the likelihood of medication-related harm post-discharge. The PRIME tool consists of eight variables drawn from clinical, medication, and psychosocial domains. Applied at the point of discharge, it provides the absolute risk of an individual older adult experiencing medication-related harm during the eight weeks after discharge from acute hospital admission. This stratification is important in order to deliver targeted interventions in resource-limited healthcare settings.

ELIGIBILITY:
Inclusion Criteria:

* Population-based cohort study that included all patients ≥18 years hospitalized in internal medicine ward at Landspitali - The National University Hospital of Iceland during the study period 1st January 2010 and 31st December 2020

Exclusion Criteria:

* Under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is Internal medicine patients in hospital settings. The cohort will include 100% of tertiary care internal medicine admissions in Iceland and 70-80% of secondary care in Iceland. The study population includes 85942 number of participants.
Sampling Method: Probability Sample
Enrollment: 85942 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of polypharmacy | Two years, one year pre-admission and one year post-admisson, 2010-2020
  Polypharmacy measured by by the number of different ATC classes of medications filled in the year preceding and year following surgery. Polypharmacy further quantified into categories of non-polypharmacy (<5), polypharmacy (5-9) and hyper-polypharmacy (≥10).

SECONDARY OUTCOMES:
Incidence of polypharmacy | Two years, one year pre-admission and one year post-admisson, 2010-2020
  Polypharmacy measured by by the number of different ATC classes of medications filled in the year preceding and year following surgery. Polypharmacy further quantified into categories of non-polypharmacy (<5), polypharmacy (5-9) and hyper-polypharmacy (≥10).
Potentially inappropriate prescribing by Beers criteria 2019 | 2010-2020
  The association of potentially inappropriate prescribing by applying Beers criteria 2019 with polypharmacy (summary score, yes/no)
Anticholinergic burden by applying the Anticholinergic burden scale | 2010-2020
  The association of anticholinergic burden by applying the Anticholinergic burden scale with polypharmacy ((summary score, yes/no)
Demographics | 2010-2020
  Gender (male, female),age (years), comorbidity based on the International Statistical Classification of Diseases, and Related Health Problems, ninth or tenth revision, ICD9/10 classification system
Comorbidity burden | 2010-2020
  The association of comorbidity burden will be described by calculating the Charlson Comorbidity Index and Elixhauser comorbidity index (summary score) with polypharmacy ((summary score, yes/no)
Drug classes | 2010-2020
  Drug classes based on ATC-codes on filled medications from the Prescription Medicines Registry and association with polypharmacy
Clinical outcomes | 2010-2020
  Mortality (short-and long-term mortality) Length of hospital stay (number of days, ≥ ten days) Readmission (number of days until readmission, readmission <30 days)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Pharmaceutical Sciences, Reykjavik, Iceland

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Derived] Jonsdottir F, Blondal AB, Gudmundsson A, Bates I, Stevenson JM, Sigurdsson MI. The association of degree of polypharmacy before and after among hospitalised internal medicine patients and clinical outcomes: a retrospective, population-based cohort study. BMJ Open. 2024 Mar 28;14(3):e078890. doi: 10.1136/bmjopen-2023-078890. PMID 38548367